CLINICAL TRIAL: NCT06391229
Title: A Brief Intervention to Enhance Supportive Parenting and Treatment Engagement Among Families Waiting for Trauma-Focused Services
Brief Title: Examine the Feasibility and Acceptability of Project Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caitlin Elizabeth Rancher, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00136524; K99HD111677 (NIH)
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Parent-Child Relations; Parenting; Child Mental Disorder
Keywords: Non-offending caregiver; Child trauma
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project Support (Experimental): All caregivers will receive the Project Support intervention over the course of 4-6 weeks.
  Interventions: Behavioral: Project Support

INTERVENTIONS:
Behavioral: Project Support — Caregivers will receive up to four, 60- to 90-minute sessions focused on teaching two parenting skills - attentive listening and comforting. Attentive listening involves providing accurate and timely responses to show interest and keep the child engaged until they are ready to end the conversation. Comforting involves using the same attentive listening skills when the child is upset or distressed. Effective mastery of the listening and comforting skills also requires caregivers to withhold any non-listening or non-comforting responses (e.g., interruptions, criticisms).
  The program is individually tailored such that caregivers with stronger skills could complete the program in less time (i.e., fewer sessions). Service providers educate caregivers about the skills, then engage in an iterative process of modeling the skills, engaging the caregivers in behavioral practice, and providing tailored, supportive feedback to help caregivers gain mastery.
  Other Names: Project Support Positive Parenting Module

SUMMARY:
In this study, the investigators will conduct a proof-of-concept pilot trial of delivering the Project Support Positive Parenting Module (Project Support) to n = 30 families waiting for trauma-focused services. Investigators hypothesize that Project Support will be feasible and acceptable as evidenced by benchmarks for recruitment, retention at post assessment, engagement, fidelity, and program satisfaction. Investigators will also explore trends on caregiver emotional support, parenting self-efficacy, and child mental health symptoms.

DETAILED DESCRIPTION:
Over two-thirds of children experience traumatic events such as child maltreatment, violence, or sudden or violent loss. Many of these children sustain significant emotional and developmental difficulties including trauma symptoms, aggression, and suicidality. Emotional support from a caregiver is theorized to buffer against the effects of trauma; however, many caregivers lack the self-efficacy and skills to effectively support their child, or struggle to apply these skills during the stressful time following trauma. Unfortunately, programs designed for caregivers following child trauma are scarce. Existing interventions are lengthy (lasting 8-20 sessions) and result in families placed on long waitlists. This proposal asserts the adverse effects of child trauma can be interrupted though a brief intervention (the Project Support Positive Parenting Module) that enhances supportive parenting - delivered via telehealth to families on waitlists for trauma-focused services. In this study, Investigators will conduct a proof-of-concept pilot trial with n = 30 families waiting for trauma-focused services. Investigators hypothesize that Project Support will be feasible and acceptable as evidenced by benchmarks for recruitment, retention at post assessment, engagement, fidelity, and program satisfaction. Investigators will also explore trends on caregiver emotional support, parenting self-efficacy, and child mental health symptoms. Long-term, this research will generate an effective intervention that addresses the needs of families affected by trauma, which can be scaled up to address other public health epidemics that impede supportive parenting and child development.

ELIGIBILITY:
Inclusion Criteria:

* Family is seeking trauma-focused services for their child as measured by their placement on the waitlist for services at the National Crime Victims Center;
* Child is between 5 - 12 years old;
* Caregiver agreed to be contacted for volunteer research opportunities;
* Caregiver and child can communicate in either English or Spanish;
* Child has been living with caregiver for at the last 6 months or longer;
* Family is able to participate in services delivered via telehealth.

Exclusion Criteria:

* Child or caregiver has a diagnosis that would impair their ability to participate in or benefit from services (e.g., traumatic brain injury, developmental disability, psychosis);
* Child is in Foster Care or Department of Social Services custody;
* The caregiver is unwilling or unable to give informed consent and/or the child is unwilling and unable to give assent.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Supportive Parenting assessed by the Alabama Parenting Questionnaire | Baseline to Post-test (6 weeks)
  Caregivers and children will complete convergent versions of the Alabama Parenting Questionnaire. Responses to this questionnaire assess several domains of parenting. Responses to items assessing supportive parenting (e.g,. "you praise your child if he/she behaves well") are made on a 5-point scale (0 = never, 1 = almost never, 2 = sometime, 3 = often, 4 = always). Responses are summed to create a total score. Higher scores of supportive parenting measured on the Alabama Parenting Questionnaire have previously been associated with lower levels of child behavior problems. This outcome measure will be assessed by comparing within-person mean levels of supportive parenting from baseline to post-test.
Parenting self-efficacy assessed by the Parenting Sense of Competence Scale | Baseline to Post-test (6 weeks)
  Caregivers will complete the parenting self-efficacy subscale of the Parenting Sense of Competence Scale. Responses to items on this questionnaire measuring self-efficacy (e.g., "If anyone can find the answer to what is troubling my child, I am the one") are made on a 6-point scale (1 = strongly disagree to 6 = strongly agree). Responses are summed to create a total score. Higher scores on the self-efficacy subscale have been associated with lower levels of child externalizing problems. This outcome measure will be assessed by comparing within-person mean levels of parenting self-efficacy from baseline to post-test.
Hopefulness assessed by the Beck Hopelessness Scale-4 | Baseline to Post-test (6 weeks)
  Caregivers will complete the Beck Hopelessness Scale-4. Responses to items on this questionnaire measuring hopelessness (e.g., "I feel the future is hopeless and that things cannot improve") are made on a 4-point scale (0 = not typical, 1 = rarely typical, 2 = typical, 3 = very typical). Responses are summed to create a total score, with higher scores indicating greater hopelessness. The Beck Hopelessness Scale-4 has demonstrated robust internal reliability, coefficient alphas = .84-.88. This outcome measure will be assessed by comparing within-person mean levels of hopelessness from baseline to post-test.

SECONDARY OUTCOMES:
Child psychological distress assessed by the Pediatric Symptom Checklist | Baseline to Post-test (6 weeks)
  Caregivers and children will complete convergent versions of the Pediatric Symptom Checklist. Responses to items on this questionnaire measuring child psychological distress (e.g., "Feels sad, unhappy") are made on a 3-point scale (0 = never, 1 = sometimes, 2 = often). Responses are summed to create a total score, with higher scores indicating greater psychological distress. Scores on the Pediatric Symptom Checklist have demonstrated convergent validity with other measures of child psychological distress. This outcome measure will be assessed by comparing within-person mean levels of child psychological distress from baseline to post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Rancher, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- National Crime Victims Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT06391229/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT06391229/ICF_002.pdf